CLINICAL TRIAL: NCT04345211
Title: The Effect of Manual Therapy, Thera-band Exercise and Walking on Age-related Lung Function and Functional Capacity
Brief Title: Manual Therapy, Thera-band Exercise and Walking
Acronym: MTBEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ID0029
Record Dates: First submitted 2020-04-05; First posted 2020-04-14 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Aging
MeSH Terms: interventions — Walking; Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group1 (G1): walking group (Active Comparator): All walks will be done immediately after the MT and TB intervention, as this has been shown to improve the synergistic effect of combining the two interventions. The walking sessions will be organized twice a week. The walking sessions will begin with a 10-minute warm-up. After warming up, you will take a continuous walk for 10-20 min, at a target intensity of 13 ("somewhat difficult") on the Borg scale. Using the Borg scale, which ranges from 6 to 20, participants will be asked to walk at an intensity of 13 (perception of "somewhat difficult" activity). Each session will be completed with a 10 minute cool down period. The objectives of Walinking will be individualized according to the level of physical condition of each participant. The walking group will include a weekly walking goal of 75 minutes.
  Interventions: Other: Group1, walking group
- Group 2 (G2): walking plus manual therapy (Active Comparator): Walking as previously described plus a self-administered manual chest therapy:
  - Neurolymphatic points pressure: Participants will be placed in a neutral position and their arms next to their bodies. They are asked to take a conscious breath. The physical therapist will apply firm, direct rotary pressure through the thumb or fingertip for 1 minute from the T1 transverse processes to the T12 transverse processes. Suboccipital decompression / mobilization, slippage of the cervical vertebral joints (anterior / posterior), myofascial release of sternocleidomastoid and trapezius, slippage of the sternoclavicular joint (anterior / posterior direction), myofascial release of intercostal muscles and paravertebral muscles (anterior rib mobilization, posterior, lateral), mobilization of the scapulothoracic joint, diaphragmatic release.
  Interventions: Other: Group 2, Walking plus manual therapy
- Group 3 (G3): walking plus thorax exercises with Theraband. (Active Comparator): Walking as previously described plus a self-administered exercises with elastic-band. The exercises will include chest and arms exercises in sitting position.
  Interventions: Other: Group 3; Walking plus exercises with Theraband
- Group 4 (G4): control group (No Intervention): Control group will do usual life and assessments as the rest of the groups.

INTERVENTIONS:
Other: Group1, walking group — The walking group includes a weekly walking goal of 75 minutes.
  Arms: Group1 (G1): walking group
Other: Group 2, Walking plus manual therapy — Walking plus self-administered thorax manual therapy
  Arms: Group 2 (G2): walking plus manual therapy
Other: Group 3; Walking plus exercises with Theraband — Walking plus thorax exercises with Theraband
  Arms: Group 3 (G3): walking plus thorax exercises with Theraband.

SUMMARY:
Worldwide, the number of older adults is expected to more than double by 2050 and more than triple by 2100, with most of the increase in developing countries. This situation has become a challenge to health professions such as physical therapy, since aging involves a gradual reduction in the capacity to adapt and an increase in vulnerability to health issues such as chronic non-communicable diseases and musculoskeletal disorders. The respiratory system, as the rest of the body, is exposed to both physiological aging and disease. According to the World Health Organization , respiratory diseases such as trachea, bronchi, or lung cancer, lower respiratory tract infections, or chronic obstructive pulmonary disease are found in the third, fifth, and sixth cause of death, respectively, among the top ten.

Therefore, bronchopulmonary and thoracic pathology constitutes an important problem for Public Health, both due to the high number of affected subjects and to their potential severity For this reason, the recommendations of the European, North American and national societies, highlight, among other aspects, the importance of the prevention of these diseases. They also insist on the need to maintain the integrity of the thoraco-abdominal anatomical elements and preventive treatment in those at risk, before symptoms appear. These recommendations together with the change of perspective that is being taken into account when treating aging have led to the fact that in the last decade more research has been started on the respiratory system in older people without respiratory problems.

The aim of this trial is to investigate whether manual therapy, elastic band exercise or walking can mitigate the effects of age-related changes in lung function in adults over 60 years old. Also whether there is a difference in effect between the different forms of therapy.

DETAILED DESCRIPTION:
Study design A 4-week program will be implemented with sessions 2 days a week, 45-60 minutes per session. It would be convenient for each group to have 30 participants each. Group1: walking group. 40 minutes walking with supervision of the physiotherapist. 2 times per week.; Group 2: walking (40 minutes) plus self-administered thorax manual therapy (20 minutes). It will be applied in group and supervised by a physiotherapist. 2 times per week.; Group 3: walking (40 minutes) plus thorax exercises with elastic-band (20 minutes). It will be applied in group and supervised by a physiotherapist. 2 times per week.;Group 4: control group will do usual life and assessments as the rest of the groups.

Oucome measures Pulmonary function: pulmonary function evaluation via forced spirometry dynamic lung volumes (forced vital capacity, FVC; forced expired volume at 1 second, FEV1). Chest wall expansion: A measuring tape is used to measure chest expansion in centimetres (cm) at two levels of the rib cage: upper chest expansion and lower chest. Exercise tolerance: 6 Six Minute Walk Test. Smoking Index. The smoking index is a unit for measuring cigarettes consumption over a long period. Musculoskeletal Pain: visual analog scale. The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations. Perception of change after treatment: Patient Global Impression of Improvement. Quality of life. Trigger points pain: by algometer. Change in thorax position: Distance between acromion-bed. Functional capacity: Sit-to-stand. Frailty: FRAIL Questionnaire. Motivation and self-efficacy: Participation motives are measured with the Exercise Motivation Index.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 60-85 years old.
* Male and female
* No history of respiratory or cardiac disease
* Currently non-smoking (> 6 months)
* Willingness to provide written consent
* Willingness to participate in and comply with study requirements

Exclusion Criteria:

* Adults over 85 years old.
* History of respiratory pathology.
* History of cardiac pathology.
* Inability to walk unaided and unassisted
* Acute pain on thoracic joint range of motion testing
* Contra-indicated for thoracic mobilisation and/or manipulation (physical screening examination)
* Inability to provide informed consent, e.g. people with a cognitive impairment, intellectual disability or mental illness

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | 4-8 week
  pulmonary function evaluation via forced spirometry dynamic lung volumes (forced vital capacity, FVC; forced expired volume at 1 second, FEV1).

SECONDARY OUTCOMES:
Chest expansion | 4-8 week
  A measuring tape is used to measure chest expansion in centimetres (cm) at two levels of the rib cage: upper chest expansion and lower chest.
Exercise tolerance | 4-8 week
  6 Six Minute Walk Test (6MWT). The object of this test is to walk as far as possible for 6 minutes. The patient will walk back and forth around the cones in a hallway and is permitted to slow down, to stop, and to rest as necessary (but resume walking as soon as able).
Smoking | 4-8 week
  The smoking index is a unit for measuring cigarettes consumption over a long period and was calculated using the following formula:
  Smoking index = Cigarettes Smoked per Day (CPD)× years of tobacco use.
  Smoking index categories were non-smoker, <400, 400-799, and ≥800. The CPD was estimated for current and former smokers. We defined heavy smoking as ≥20 CPD and mild smoking as <20 CPD.
  The smoking index is a unit for measuring cigarettes consumption over a long period and was calculated using the following formula:
  Smoking index = Cigarettes Smoked per Day (CPD)× years of tobacco use.
  Smoking index categories were non-smoker, <400, 400-799, and ≥800. The CPD was estimated for current and former smokers. We defined heavy smoking as ≥20 CPD and mild smoking as <20 CPD.
Musculoskeletal Pain | 4-8 week
  visual analog scale (VAS). The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations.
Perception of change after treatment | 4-8 week
  By Patient Global Impression of Improvement (PGIC).
Perception of Quality of life | 4-8 week
  By SF-8 scale. The SF-8 consists of 8 items comprising 8 dimensions (Bodily Pain, Perceptions, Mental Health, Physical Function, Role-physical, Role-emotional, Social Function, and Vitality).
  To assess each dimension, items are aggregated into a score ranging from 0 to 100; being higher scores indicators of good health.
Trigger points pain | 4-8 week
  By algometer. Pressure was applied perpendicular to the skin, at a speed of 30kPa/s. Three measurements with 1 minute between measurements were averaged.
Change in thorax position | 4-8 week
  Distance between acromion-bed.To assess the position of the upper trunk, the length of the pectoralis minor in the supine position is evaluated by measuring the distance between the posterior edge of the acromion and the stretcher while the patients remain in that position.
Functional capacity | 4-8 week
  By Sit-to-stand test. Participants sit in a 43 cm tall armless chair (Fig. 1) as quickly as possible 5 times. Participants cross their arms over their chest and are instructed to fully stand up and make firm contact when sitting. Time begins with the "go" command and ends when participants sit down after the fifth stand-up.
Frailty | 4-8 week
  By FRAIL Questionnaire. The FRAIL scale are short 5-question assessment of fatigue, resistance, aerobic capacity, illnesses, and loss of weight, classified the patients into 3 categories: robust (score = 0), prefrail (score = 1-2), and frail (score = 3-5).
Motivation and self-efficacy | 4-8 week
  Participation motives are measured with the Exercise Motivation Index. The questionnaire consists of 15 statements followed by a five-point rating scale for each statement, ranging from 0 (not important) to 4 (extremely important). Although the authors found that the index was valid and reliable, they advise that further validation be made. Three subscores (0-4) were calculated by summing the scores for physical, psychological, and social motivation and dividing them by the number of statements for each area (Stenström, 1997; Klompstra, 2015) Cronbach's alpha was 0.889.
Screening sarcopenia | 4-8 week
  Screening sarcopenia: SARC-F. There are 5 components of SARC-F questionnaire: strength, assistance with walking, rise from a chair, climb stairs, and fall. The SARC-F scores range from 0 to 10, with 0 to 2 points for each component. A score ≥4 is predictive of sarcopenia and poor outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma V Espí-López, Dr, Principal Investigator — Faculty of Physiotherapy. University of Valencia
Locations (1):
- Gemma Espí, Valencia, Spain